CLINICAL TRIAL: NCT00615875
Title: Naproxen for Acute Pain After Surgery: A Randomized, Placebo-Controlled Trial
Acronym: NAPS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Tuan Dinh, Pharmacy Department, St. Joseph's Healthcare Hamilton
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 07-2936
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Last update posted 2008-02-14 (Estimated); Status verified 2008-01

CONDITIONS: Pain, Postoperative
Keywords: naproxen; acute pain; postoperative pain; thoracic surgery; head and neck surgery; opiate sparing
MeSH Terms: conditions — Pain, Postoperative; Acute Pain | interventions — Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: naproxen
- P (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: naproxen — opaque pale orange suspension: 20mL q12h x 4 doses mixed in juice.
  Other Names: Naprosyn suspension (Roche)
  Arms: A
Drug: placebo — opaque pale orange suspension: 20mL q12h x 4 doses mixed in juice
  Arms: P

SUMMARY:
The purpose of this study is to determine whether using an additional 48 hours of oral naproxen, after other post-operative pain medications have been stopped, will be effective in reducing opiate pain medication requirements and contribute to improved pain management.

DETAILED DESCRIPTION:
At St. Joseph's Healthcare Hamilton, the Acute Pain Service (APS) is responsible for the immediate post-operative pain management of many surgical inpatients. While cared for by APS, the patient receives multimodal analgesia, including adjunctive medications (acetaminophen and naproxen/ketorolac) scheduled around the clock. When APS discontinues the epidural/pain pump, all adjunctive medications are discontinued and the patient is usually started on 'as needed' opiate or combination opiate (i.e. Tylenol#3) medications. On occasion, APS will write an order for an additional 48 hours of naproxen, but this practice has not been formally evaluated at this site. This randomized, placebo-controlled study proposes to evaluate this bridging strategy to see if regularly scheduled naproxen after discontinuation of other post-operative medications will affect the daily doses of opiate pain medications used, side effects of those opiate medications and pain scores of patients.

ELIGIBILITY:
Inclusion Criteria:

* undergone Head & Neck and Thoracic surgery
* admitted to Chest, Head and Neck or Step-Down at St. Joseph's Healthcare
* pain management by APS (epidural/pain pump) including naproxen/ketorolac
* able to take oral medications (by mouth, feeding tube or NG tube)
* reasonably able to communicate in English and provide consent

Exclusion Criteria:

* pre-existing chronic pain (morphine equivalent doses over 200mg/day in 5 days previous to surgery)
* recovering from cardiac, urological, orthopedic, laparoscopic or ambulatory surgery
* chronic NSAID therapy (daily for more than 3 weeks or high dose (over 81mg) ASA at least 4 days/week for more than 3 weeks)
* pregnancy, diagnosis of sepsis, history of stroke or transient ischemic attack, CHF (NYHA 3 or 4), allergy or contraindication to NSAIDS as defined by APS protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-05 (Estimated); Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
cumulative opiate dose administered, as recorded on the computerized medication administration record (CMAR) | daily

SECONDARY OUTCOMES:
patient reported pain scores | at least three times daily
side effects of study medication and opiate analgesia | at least three times daily

CONTACTS AND LOCATIONS:
Overall Officials: Tuan Dinh, RPh, Principal Investigator — St. Joseph's Healthcare Hamilton
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Starck PL, Sherwood GD, Adams-McNeill J, Thomas EJ. Identifying and addressing medical errors in pain mismanagement. Jt Comm J Qual Improv. 2001 Apr;27(4):191-9. doi: 10.1016/s1070-3241(01)27017-5. PMID 11293836
- [Background] Apfelbaum JL, Chen C, Mehta SS, Gan TJ. Postoperative pain experience: results from a national survey suggest postoperative pain continues to be undermanaged. Anesth Analg. 2003 Aug;97(2):534-540. doi: 10.1213/01.ANE.0000068822.10113.9E. PMID 12873949
- [Background] Callesen T, Bech K, Kehlet H. Prospective study of chronic pain after groin hernia repair. Br J Surg. 1999 Dec;86(12):1528-31. doi: 10.1046/j.1365-2168.1999.01320.x. PMID 10594500
- [Background] Joshi GP. Multimodal analgesia techniques and postoperative rehabilitation. Anesthesiol Clin North Am. 2005 Mar;23(1):185-202. doi: 10.1016/j.atc.2004.11.010. PMID 15763418
- [Background] Hartrick CT. Multimodal postoperative pain management. Am J Health Syst Pharm. 2004 Apr;61 Suppl 1:S4-10. doi: 10.1093/ajhp/61.suppl_1.S4. PMID 15119755
- [Background] Cepeda MS, Carr DB, Miranda N, Diaz A, Silva C, Morales O. Comparison of morphine, ketorolac, and their combination for postoperative pain: results from a large, randomized, double-blind trial. Anesthesiology. 2005 Dec;103(6):1225-32. doi: 10.1097/00000542-200512000-00018. PMID 16306736
- [Background] Richy F, Bruyere O, Ethgen O, Rabenda V, Bouvenot G, Audran M, Herrero-Beaumont G, Moore A, Eliakim R, Haim M, Reginster JY. Time dependent risk of gastrointestinal complications induced by non-steroidal anti-inflammatory drug use: a consensus statement using a meta-analytic approach. Ann Rheum Dis. 2004 Jul;63(7):759-66. doi: 10.1136/ard.2003.015925. PMID 15194568